CLINICAL TRIAL: NCT03058978
Title: Assessing Ovarian Function During Prolonged Implant Use
Status: Completed | Type: Observational
Sponsor: Planned Parenthood of the St. Louis Region and Southwest Missouri (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 201612108
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Etonogestrel Implant — Ovarian function will be assessed with weekly serum progesterone levels. Participants will undergo weekly venipuncture for a total of four draws over a 30 day period. Participants will also complete a bleeding diary to assess daily bleeding patterns for the 30 day study period.
  Other Names: Subdermal arm implant

SUMMARY:
The study will evaluate how the ovaries may be functioning while using the the Implanon®/Nexplanon® during the three years beyond the FDA approved duration. Ovarian function will be assessed with weekly serum progesterone levels. Participants will undergo weekly venipuncture for a total of four draws. Participants will be followed for 30 days.

DETAILED DESCRIPTION:
This prospective cohort will evaluate the ovarian function of 210 ENG users during the three years beyond the FDA approved duration. Participants enrolled in the current study, EPIC (Evaluating the Prolonged Use of IUD and Implant for Contraception, NCT02267616), will be contacted via telephone, screened and scheduled to enroll in person. After the signed consent is obtained participants will be asked to complete a brief questionnaire on demographic information and bleeding patterns. Participants will undergo a blood draw to assess serum etonogestrel and serum progesterone levels.

Follow up visits will include a weekly blood draw for three weeks to assess serum progesterone levels. Participants will also complete a bleeding diary to assess daily bleeding patterns for the 30 day study period.

The investigators will enroll participants at seven time points; at method expiration (3 years of use), and in six-month intervals through six years of use.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the prospective EPIC Prolonged Use Study
* 18-45 years of age
* At expiration or beyond the end of the FDA-approved duration of use of the etonogestrel-releasing subdermal implant (ENG implant =3 years)
* Ability to consent in English
* Willing and able to complete required follow-up for the study.

Exclusion Criteria:

* Have history of female sterilization procedure
* Desire for conception in the next 12 months
* Had their ENG implant removed

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: ENG implants users who are at expiration or beyond the end of the FDA-approved duration of use of the etonogestrel-releasing subdermal implant (ENG implant =3 years)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Ovulatory function by body mass index, (kg/m^2) | 30 day period
  Comparisons of serum progesterone levels between BMI (kg/m^2) categories will be made using ANOVA or Kruskal-WIllis depending on the normality of distribution.

SECONDARY OUTCOMES:
Measure number of bleeding days while using the implant during the 30 day study period | 30 day period
  Participant self-report, daily bleeding diary

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McNicholas, DO, MSCI, Principal Investigator — Planned Parenthood of the St. Louis Region and Southwest Missouri
Locations (2):
- United States (2):
  - Planned Parenthood of the St. Louis Region and Southwest Missouri, St Louis, Missouri
  - Washington University in St Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No